CLINICAL TRIAL: NCT07063511
Title: A Prospective Clinical Trial Evaluating the Safety and Efficacy of Concurrently Layering Hyaluronic Acid Fillers in Different Tissue Planes During Facial Aesthetic Treatments
Brief Title: Pan-Facial Layering of Hyaluronic Acid Filler
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAL-2025-LAYER-62
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Aesthetic
Keywords: Hyaluronic Acid; Fillers; Facial Assessment; Multilayering Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Restylane Injectables (Other): Thirty (30) adult (> 18 years) participants, including fifteen (15) participants with a primary deficit of the midface, and fifteen (15) participants with a primary deficit of the lower face (chin, lips) as assessed by the Treating Investigator. Primary deficit is defined as facial third requiring more intense treatment or volumes of HA.
  Interventions: Device: Restylane Injectables

INTERVENTIONS:
Device: Restylane Injectables — Participants will receive multilayering treatment (i.e., one product will be placed deep and one in a more superficial plane) in area of primary deficit (i.e., the midface or lower face), in isolation or combination with other treatment areas.

SUMMARY:
Recent advancements in anatomical studies have enabled a more sophisticated approach to treating patients with facial aesthetic concerns with hyaluronic acid (HA) fillers. For instance, volumizing a specific area of concern may be warranted, but it is essential to understand how the underlying patient anatomy is continuing to laxity and hollowness.

Varying manufacturing technology have offered a range of HA fillers with different physical and chemical properties adapted to different indications, each one tailored to provide a slightly different outcome based on the needs of the patient.

Given these advances in the medical aesthetic field, investigators and clinicians are seeking to develop a new methodology for providing patients with a more tailored and personalized treatment approach. This methodology includes using a pan-facial, multilayering treatment technique that can be employed by injectors once experience is gained with standard techniques.

The goal of this study is to assess the efficacy and safety of layering HA from the Restylane line of soft tissue products to create a more harmonious and complete aesthetics results.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily sign and date an informed consent, approved by an independent ethics committee, prior to the initiation of any screening or study-specific procedures.
2. Participants must be adult male or female, at least 18 years old.
3. Participants must be willing and able to comply with procedures required in the protocol.
4. Participants must be in good health as per investigator's judgment based on medical history.
5. Participants must not have uncontrolled systemic disease.
6. Participants do not present with or have a history of any medical condition that may place the participant at increased risk following exposure to hyaluronic acid or interfere with the study evaluation, including:

   * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
   * History of facial nerve palsy
   * Infection or dermatological condition at the treatment injection sites
   * Marked facial dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, or excessively photodamaged skin
7. Participants do not have history of clinically significant medical conditions or any other reason that the investigator determines would interfere with the participants participation in this study or would make the participant an unsuitable candidate to receive the study medical device.
8. Participants do not have history of an allergic reaction or significant sensitivity to constituents of the study medical device (or its excipients), including local anaesthetic agents found in the product (Lidocaine).
9. Participants must not have tattoos, jewellery, or clothing which obscure the treatment area and cannot be removed.
10. Participants do not have anticipated need for surgery or overnight hospitalization during the study.
11. Participants do not have history of surgical procedures in the face, including any lifting procedure (e.g., facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery).
12. Participants have not had, in the last 2 years, facial treatment with semi- permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
13. Participant has not received treatment with energy-based devices in the last 6 months.
14. Participant has not received soft tissue filler within the last 12 month in the face.
15. Female participants of child-bearing potential must have a negative urine pregnancy test prior to any dose of study drug.
16. Female participants of childbearing potential must practice at least 1 protocol-specified method of birth control that is effective from Baseline through at least 30 days after the last dose or until the end of study, whichever is longer. Female participants of non-childbearing potential do not need to use birth control.
17. Female participants that are not pregnant or breastfeeding and are not considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of study medical device or until the end of study, whichever is longer.
18. Participants must not have been treated with any investigational product within 30 days prior to the first dose of study medical device or is currently enrolled in another clinical study
19. Participants must not be presenting with porphyria.
20. Participants must not present with active disease, such as inflammation, infection or tumours, cold sores in or near the intended treatment sites.
21. Participants must not have bleeding disorders or take thrombolytics or anticoagulants.
22. Participants agree to abstain from taking any over the counter NSAIDs at least two weeks prior to any treatment administration (e.g. Advil)
23. Participants must not have need to take immunosuppressants.

Exclusion Criteria:

1. Participants with known active COVID infection within 14 days of baseline treatment.
2. Participants has a history of cystic acne.
3. Participant has had or is planning to have dental procedures, including teeth cleaning procedures at least 2 weeks before or after any scheduled treatment administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) related to multilayering treatment technique | Baseline to Week 24
  Safety of multilayering treatment technique will be determined by the frequency and severity of adverse events (AEs): a. physician-reported and b. participant-reported.
Evaluate the efficacy of concurrently layering hyaluronic acid fillers in different tissue planes during facial aesthetic treatments in the same region at different depths | Baseline to Week 24
  The efficacy of multilayering treatment technique will be determined by the frequency of participants having at least "improved" (e.g., "improved", "much improved" or "very much improved") on the Global Aesthetics Improvement Scale (GAIS), a 5-point scale, categorized as "worse", "no change", "improved", "much improved", and "very much improved", as graded by a blinded evaluator.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, Principal Investigator — Erevan Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No